CLINICAL TRIAL: NCT02504723
Title: Carvedilol Plus Endoscopic Cyanoacrylate Injection Versus Endoscopic Cyanoacrylate Injection for Secondary Prophylaxis of Gastric Variceal Bleeding
Brief Title: Carvedilol as an Adjunct to Endoscopic Cyanoacrylate Injection for Secondary Prophylaxis of Gastric Variceal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Wen-Chi Chen, MD, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS11-CT10-11
Record Dates: First submitted 2015-07-18; First posted 2015-07-22 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Esophageal and Gastric Varices
Keywords: Gastric varices; cyanoacrylate; carvedilol
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Carvedilol; Cyanoacrylates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyanoacrylate injection plus carvedilol (Experimental): The patients undergo repeated endoscopic cyanoacrylate injection every 3-4 weeks until obturation of gastric varices. Oral carvedilol is administrated during the whole study period, starting at 6.25 mg daily and increased until the maximum tolerated dose.
  Interventions: Drug: carvedilol; Drug: cyanoacrylate
- Cyanoacrylate injection (Active Comparator): The patients undergo repeated endoscopic cyanoacrylate injection every 3-4 weeks until obturation of gastric varices.
  Interventions: Drug: cyanoacrylate

INTERVENTIONS:
Drug: carvedilol — Oral carvedilol is started after randomization at an initial dose of 6.25 mg daily. Doses are increased every 3 days during the admission or every 7 days in the out-patient clinics until the maximum tolerated dose was achieved or up to 25 mg daily, aiming at reducing resting pulse rate by 25 percent but not below 55 beats per minute with systolic blood pressure >90 mm Hg.
  Arms: Cyanoacrylate injection plus carvedilol
Drug: cyanoacrylate — The patients undergo repeated endoscopic cyanoacrylate injection every 3-4 weeks until obturation of gastric varices.

SUMMARY:
Gastric variceal obturation is the current endoscopic therapy of choice for gastric variceal bleeding but is associated with a high rebleeding rate. Carvedilol is a potent non-selective β-blocker. The role of carvedilol in the prevention of recurrent gastric variceal bleeding is not studied. This study aimed at evaluating the efficacy of carvedilol as an adjunct to gastric variceal obturation in the secondary prophylaxis of gastric variceal bleeding.

DETAILED DESCRIPTION:
Gastric variceal bleeding is a lethal complication of portal hypertension. The rebleeding rate ranged between 30% to 50% in patients after initial hemostasis. Endoscopic cyanoacrylate injection is currently the choice of endoscopic therapy of acute gastric variceal bleeding and prevention of recurrent bleeding. However, the rebleeding rate is still high in the patients undergoing repeated endoscopic cyanoacrylate injection.

Non-selective β-blockers are frequently used for the secondary prophylaxis of variceal bleeding. In the case of esophageal varices, combination of non-selective β-blockers and endoscopic therapy significantly lowers the rebleeding rate compared with endoscopic therapy alone. However, propranolol failed to decrease the rebleeding rate as an adjunct to endoscopic cyanoacrylate injection and was associated with a higher incidence of adverse effects in gastric variceal bleeding patients. A more potent non-selective β-blocker than propranolol might further decrease portal pressure and decrease the rebleeding rate.

Carvedilol is a potent non-selective β-blocker with both beta and alpha-1 blocker effect. It significantly lowers portal pressure even in propranolol non-responders. However, it is unclear weather carvedilol will play a role in the prevention of recurrent gastric variceal bleeding. The investigators conducted a randomized controlled trial to compare the efficacy of carvedilol combined with endoscopic cyanoacrylate injection with endoscopic cyanoacrylate injection alone in secondary prophylaxis of gastric variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 to 80 years
* Cirrhotic patients with acute gastric variceal bleeding proven by an endoscopy within 24 h of bleeding
* Stable hemodynamic condition for at least 3 days after cyanoacrylate injection

Exclusion Criteria:

* Previous treatment of gastric varices, including endoscopic therapy, transjugular intrahepatic porto-systemic shunt, or surgery
* Contraindications to non-selective beta-blockers or cyanoacrylate injection
* Serum total bilirubin >10 mg/dL
* Grade III/IV hepatic encephalopathy
* Hepato-renal syndrome
* Severe heart failure (NYHA Fc III/IV)
* Chronic kidney disease under renal replacement therapy
* Refractory ascites
* Malignancy other than hepatocellular carcinoma
* Pregnancy
* Pacemaker use
* Refusal to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chi Chen, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Chen WC, Hsin IF, Chen PH, Hsu PI, Wang YP, Cheng JS, Lin HS, Hou MC, Lee FY. Addition of Carvedilol to Gastric Variceal Obturation Does Not Decrease Recurrence of Gastric Variceal Bleeding in Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2019 Oct;17(11):2356-2363.e2. doi: 10.1016/j.cgh.2019.02.021. Epub 2019 Feb 14. PMID 30772583

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyanoacrylate Injection Plus Carvedilol | Cyanoacrylate Injection
Started | 60 | 61
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyanoacrylate Injection Plus Carvedilol | Cyanoacrylate Injection | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.52 (10.87) | 56.26 (12.08) | 56.39 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 41 | 41 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rebleeding From Gastric Varices
Description: Rebleeding from gastric varices during the follow-up period
Time Frame: Within 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cyanoacrylate Injection Plus Carvedilol | Cyanoacrylate Injection
Number analyzed (Participants) | 60 | 61
Participants | 14 | 21

2. Secondary Outcome: All Upper Gastrointestinal Bleeding
Description: All upper gastrointestinal bleeding during the follow-up period
Time Frame: Within 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cyanoacrylate Injection Plus Carvedilol | Cyanoacrylate Injection
Number analyzed (Participants) | 60 | 61
Participants | 17 | 29

3. Secondary Outcome: All Cause Mortality or Liver Transplantation
Description: All cause mortality or liver transplantation during the study period
Time Frame: Within 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cyanoacrylate Injection Plus Carvedilol | Cyanoacrylate Injection
Number analyzed (Participants) | 60 | 61
Participants | 13 | 20

4. Secondary Outcome: All Adverse Effects
Description: All adverse effects during the study period
Time Frame: Within 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cyanoacrylate Injection Plus Carvedilol | Cyanoacrylate Injection
Number analyzed (Participants) | 60 | 61
Participants | 32 | 9

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Cyanoacrylate Injection Plus Carvedilol | Cyanoacrylate Injection
All-Cause Mortality (participants affected / at risk) | 12/60 | 19/61
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 32/60 | 9/61
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyanoacrylate Injection Plus Carvedilol (N=60) | Cyanoacrylate Injection (N=61)
dizziness (General disorders) | 11 (11) | 1 (1)
weakness (General disorders) | 2 (2) | 1 (1)
hypotension (General disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
abdominal pain (General disorders) | 1 (1) | 2 (2)
insomnia (General disorders) | 2 (2) | 1 (1)
chronic cough (General disorders) | 1 (1) | 0 (0)
dyspnea on exertion (General disorders) | 8 (8) | 0 (0)
poor gastric ulcer healing (Gastrointestinal disorders) | 1 (1) | 2 (2)
dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
recurrent bacteremia (Infections and infestations) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02504723/Prot_SAP_001.pdf